CLINICAL TRIAL: NCT05424523
Title: A Retrospective Multicenter Study for Assessment of the Effectiveness and Safety of Omalizumab in Children With Allergic Asthma in a Real-world Setting in China
Brief Title: Effectiveness and Safety of Omalizumab in Children With Allergic Asthma.
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CIGE025BCN01
Record Dates: First submitted 2022-06-15; First posted 2022-06-21 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Allergic Asthma
Keywords: Omalizumab,; allergic asthma,; children,; real-world study
MeSH Terms: interventions — Omalizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Omalizumab: Patients with confirmed diagnosis of allergic asthma, who were prescribed omalizumab
  Interventions: Drug: Omalizumab

INTERVENTIONS:
Drug: Omalizumab — Patients with confirmed diagnosis of allergic asthma, who were prescribed omalizumab

SUMMARY:
The study was the non-interventional, retrospective study aimed to assess the effectiveness and safety of omalizumab in children with allergic asthma in China, and described patient profiles and treatment patterns of omalizumab in real-world practice.

DETAILED DESCRIPTION:
This non-interventional, retrospective study aimed to assess the effectiveness and safety of omalizumab in children with allergic asthma in China, and described patient profiles and treatment patterns of omalizumab in real-world practice. This study was designed to use secondary data from medical charts of 25 hospitals. Medical records were reviewed to collect information such as demographics, clinical characteristics, treatment patterns, effectiveness, and AEs for retrospective analysis. Patients with allergic asthma aged 6 -<12 years treated with omalizumab from July 6, 2018 to September 30, 2020 were identified for medical chart extraction.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 6 -<12 years
* Diagnosed with allergic asthma and could be treated using omalizumab. Comorbidities included allergic rhinitis, atopic dermatitis, nasal polyp, chronic urticaria, and food allergy
* Received omalizumab during the identification period
* Had at least one documented follow-up data after omalizumab treatment
* Provided informed consent if required by ethics committee (EC) of hospital

Exclusion Criteria:

* Current participation in a clinical trial of any investigational treatment

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients with allergic asthma treated with omalizumab from July 6, 2018 to September 30, 2020 were identified for medical chart extraction
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2021-06-28 (Actual); Study Completion 2021-06-28 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who responded to omalizumab | After 4-6 months of treatment (Between July 6, 2018 to September 30, 2020)
  The responders were defined as patients with:
  1. Investigator's Global Evaluation of Treatment Effectiveness (GETE) are Excellent or Good; or
  2. C-ACT2 improvement ≥3 points before and after omalizumab treatment

SECONDARY OUTCOMES:
Number of adverse events and serious adverse events | Throughout the study, approximately 2 years
  To evaluate safety of omalizumab among children with allergic asthma in China.
Proportion of patients with positive investigator's Global Evaluation of Treatment Effectiveness (GETE) | After 4-6 months of treatment (Between July 6, 2018 to September 30, 2020)
  Positive investigator's GETE is defined as restrospectively evaluated GETE are Excellent or Good.
Change from baseline in moderate-to-severe Asthma exacerbation | Baseline, after 4-6 months of treatment (Between July 6, 2018 to September 30, 2020)
  Moderate-to-severe asthma exacerbation is defined as worsening of asthma symptoms requiring doubling of baseline ICS dose and/or treatment with rescue systemic corticosteroids for ≥ 3 days.
Change from baseline in severe Asthma exacerbation | Baseline, after 4-6 months of treatment (Between July 6, 2018 to September 30, 2020)
  Severe asthma exacerbation is defined as requiring ER admission
  /hospitalization/ICU admission/mechanical ventilation with systemic corticosteroids for ≥ 3 days.
Average change from baseline in daily inhaled corticosteroids (ICS) dose | Baseline, after 4-6 months of treatment (Between July 6, 2018 to September 30, 2020)
  The dosage of inhaled corticosteroids (ICS) was reported to evaluate the effectiveness of omalizumab among children aged 6 -<12 years with allergic asthma in China.
Average change from baseline in daily oral corticosteroids (OCS) dose | Baseline, after 4-6 months of treatment (Between July 6, 2018 to September 30, 2020)
  The dosage of oral corticosteroids (OCS) was reported to evaluate the effectiveness of omalizumab among children aged 6 -<12 years with allergic asthma in China.
Percentage of patients that successfully stopped Oral Corticosteroids | After 4-6 months of treatment (Between July 6, 2018 to September 30, 2020)
  Percentage of patients that successfully stopped Oral Corticosteroids after 4 to 6 months of treatment were reported
Change from baseline in Lung function using Forced Expiratory Volume in 1 Second (FEV1) | Baseline, after 4-6 months of treatment (Between July 6, 2018 to September 30, 2020)
  Lung function was assessed using Forced Expiratory Volume in 1 Second (FEV1) to evaluate the effectiveness of omalizumab among children aged 6 -<12 years with allergic asthma in China. FEV1 is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation.
Change from baseline in FEV1% pred | Baseline, after 4-6 months of treatment (Between July 6, 2018 to September 30, 2020)
  Ratio of patient's actual results compared to predicted normal values, expressed as a percentage.
Change from baseline in FEV1/FVC | Baseline, after 4-6 months of treatment (Between July 6, 2018 to September 30, 2020)
  The FEV1/FVC ratio indicates how much air you can forcefully exhale.
Change from baseline in Peak Expiratory Flow (PEF) | Baseline, after 4-6 months of treatment (Between July 6, 2018 to September 30, 2020)
  Peak Expiratory Flow (PEF) is an objective measure of how well the lungs are functioning and can measure airway narrowing.
Change from baseline in Maximal mid-expiratory flow (MMEF) | Baseline, after 4-6 months of treatment (Between July 6, 2018 to September 30, 2020)
  Maximal mid-expiratory flow (MMEF) is a spirometric parameter reflecting airflow of large and small airways.
Number of patients who received the recommended dosage instructions during the identification period | Throughout the study, approximately 2 years
  To describe the treatment pattern of omalizumab among children with allergic asthma in China.
Median time to discontinuation of the treatment | Throughout the study, approximately 2 years
  To describe the treatment pattern of Xolair among children with allergic asthma in China.
Percentage of patients using Omalizumab for more than 4, 16, 24 and 52 weeks | Week 4, 16, 24 and 52 (Between July 6, 2018 to September 30, 2020)
  To describe the treatment pattern of omalizumab among children with allergic asthma in China.
Number of patients who discontinued omalizumab | Throughout the study, approximately 2 years
  To describe the treatment pattern of omalizumab among children with allergic asthma in China.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, East Hanover, New Jersey, United States

REFERENCES:
- See also: Results for CIGE025BCN01 from the Novartis Clinical Trials Results Database — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17947